CLINICAL TRIAL: NCT01006915
Title: Surgical Peripheral Nerve Decompression for the Treatment of Diabetic Neuropathy in the Foot
Brief Title: Surgical Decompression for Diabetic Neuropathy in the Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy J. Best Medicine Professional Corporation (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPNPSI-1
Record Dates: First submitted 2009-10-16; First posted 2009-11-03 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Diabetic Polyneuropathy
Keywords: Diabetic sensorimotor polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical decompression (Experimental): Surgical decompression of the common peroneal, tibial, and deep peroneal nerves
  Interventions: Procedure: Surgery
- Standard medical care (No Intervention): Standard diabetic care and medical care provided for diabetic sensorimotor polyneuropathy

INTERVENTIONS:
Procedure: Surgery — Surgical decompression of the common peroneal, tibial, and deep peroneal nerves
  Arms: Surgical decompression

SUMMARY:
The purpose of the study is to determine whether or not surgical decompression of the common peroneal, tibial, and deep peroneal nerves in the legs of persons with diabetic peripheral neuropathy is effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Presence of Type 1 or 2 diabetes mellitus (fasting plasma glucose > 7 mmol/L or casual plasma glucose > 11.1 mmol/L and symptoms of diabetes or a 2hr plasma glucose in a 75g oral glucose tolerance test > 11.1 mmol/L)
* Symptoms of paresthesias (including burning pain) or numbness present symmetrically in both feet, determined to be on a peripheral nerve basis
* Total Neuropathy score of ≥ 2 based on symptoms, signs, and nerve conduction study abnormality
* Average pain on Likert scale (range 0 - 10) ≥5
* Good diabetic control with Hgb A1C < 8
* Presence of Tinel's sign at the Tarsal Tunnel
* Possession of valid Ontario Hospital Insurance Plan (OHIP) coverage

Exclusion Criteria:

* Other types of diabetes mellitus (gestational, drug-induced, etc.)
* Other cause of neuropathy than diabetes such as vasculitis, amyloidosis, toxic neuropathy, HIV, renal failure, alcohol abuse, etc. Pure entrapment neuropathy without evidence of DSP
* Symptomatic lumbosacral spine disease
* Symptomatic lower extremity vascular disease
* Previous foot ulceration or amputation. Other contraindications to surgery such as significant ankle edema, venous stasis, morbid obesity, or previous surgery/injury which would be incompatible with appropriate wound healing
* History of Peripheral Arterial Disease
* HbA1c > 8.0 - Adults lacking capacity to consent, pregnant women, prisoners, non-English speakers who require an interpreter, and those unwilling or unable to participate in the full study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-03; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To determine if lower extremity nerve decompression in patients suffering from symptomatic diabetic peripheral neuropathy significantly alleviates pain. | 0,3,6, and 12 months

SECONDARY OUTCOMES:
Neuropathic Symptoms as measured by the Total Neuropathy Score (TNS) | 0,3,6, and 12 months
Signs of peripheral neuropathy - two-point discriminations and pressure thresholds, vibration sensibility | 0 and 12 months
Nerve Conduction Velocity | 0 and 12 months
Quality of Life | 0,3,6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Best, MD, MSc, Principal Investigator — Northern Ontario School of Medicine; Sante Fratesi, MD, MSc, Study Director — Northern Ontario School of Medicine
Locations (1):
- Sault Area Hospital, Sault Ste. Marie, Ontario, Canada